CLINICAL TRIAL: NCT02283736
Title: Efficacy of Oral Probiotic Administration in Clinical, Immunological and Microbiological Parameters of Patients With Chronic Periodontitis Treated With Non Surgical Periodontal Treatment.
Brief Title: Efficacy of Oral Probiotic Administration in Patients With Chronic Periodontitis
Acronym: probiotic
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jorge Gamonal (Other)
Responsible Party: Sponsor-Investigator, Jorge Gamonal, Professor, University of Chile
Organization: University of Chile (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FONDECYT 1130570
Record Dates: First submitted 2014-11-01; First posted 2014-11-05 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: -Chronic Periodontitis
Keywords: Chronic periodontitis; Probiotics; Non- surgical treatment
MeSH Terms: conditions — Chronic Periodontitis | interventions — Dimethyl Sulfoxide; Periodontal Index

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Periodontal treatment, Probitic (Experimental): Periodontal treatment (scaling and root planning) and one tablet containing Lactobacillus rhamnosus SP1 per day during 3 months.
  Interventions: Other: Lactobacillus rhamnosus SP1; Procedure: Periodontal treatment
- Periodontal treatment, talc powder tab (Placebo Comparator): Periodontal treatment (scaling and root planning) and one tablet containing talc powder per day during 3 months
  Interventions: Other: Talc powder; Procedure: Periodontal treatment

INTERVENTIONS:
Other: Lactobacillus rhamnosus SP1 — Tablet containing Lactobacillus rhamnosus SP1
  Arms: Periodontal treatment, Probitic
Other: Talc powder — Tablet containing talc powder
  Arms: Periodontal treatment, talc powder tab
Procedure: Periodontal treatment — Scaling and root planning

SUMMARY:
The aim of this randomized placebo- controlled clinical trial is to evaluate the effects of Lactobacillus rhamnosus SP1- containing probiotic tablets as an adjunct to scaling and root planning (SRP).

Material and methods: Thirty six chronic periodontitis patients will be recruited and monitored clinically, immunologically and microbiologically at baseline, 3 and 6 months after therapy. All patients will receive scaling and root planning and randomly will be assigned over an experimental (SRP + probiotic, n=18) or control (SRP + placebo, n=18) group. The tablets will be used once per day during 3 months.

ELIGIBILITY:
Inclusion Criteria:

* ≥14 natural teeth, excluding third molars
* ≥10 posterior teeth
* ≥35 years old
* ≥ 5 teeth with periodontal sites with probing depths ≥5mm, clinical attachment loss ≥3mm
* Bleeding on probing ≥20% of sites
* Extensive bone loss determined radiographically

Exclusion Criteria:

* Periodontal treatment before the time of examination
* Systemic illness
* Pregnancy
* Anticoagulant, antibiotics and non- steroid anti- inflammatory therapy in the 6-month period before the study

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Differences of at least 1mm between groups for clinical attachment level changes | baseline, 3, 6 months

SECONDARY OUTCOMES:
Differences between groups for probing depth changes | baseline, 3, 6 month
Differences between groups for bleeding on probing changes | baseline, 3, 6 months
Differences between groups for plaque index changes | baseline, 3, 6 months
Differences between groups for levels of Interleukin (IL)-17, IL-21, Transforming Growth Factor (TGF)- beta, IL-10, RANKL changes in gingival crevicular fluid | baseline, 3, 6 months
Differences between groups for levels of periodontal pathogens changes | baseline, 3, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Gamonal, Professor, Principal Investigator — Faculty of Dentistry of University of Chile
Locations (1):
- Faculty of Dentistry of University of Chile, Santiago, Santiago Metropolitan, Chile